CLINICAL TRIAL: NCT03610984
Title: Cohort Study of Patients With Type 1 Diabetes：Clarifing the Underlying Hereditary and Autoimmune Pathogenic Factors
Brief Title: Cohort Study of Patients With Type 1 Diabetes
Status: Completed | Type: Observational
Sponsor: Second Xiangya Hospital of Central South University (Other)
Responsible Party: Principal Investigator, Zhiguang Zhou, Professor,Institute of Metabolism and Endocrinology, The Second Xiangya Hospital and the Diabetes Center, Key Laboratory of Diabetes Immunology, Ministry of Education, Central South University, National Clinical Research Center for Metabolic Diseases., Second Xiangya Hospital of Central South University
Other Study IDs: T1D Cohort Study
Record Dates: First submitted 2018-05-11; First posted 2018-08-02 (Actual); Last update posted 2022-07-06 (Actual); Status verified 2022-07

CONDITIONS: Type 1 Diabetes Mellitus; Structured Education
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Intensive structured education group: Regular outpatient visit in every 3 months to these patients. The glucose control and diabetes complication screening will be evaluated in visit. Patients will also be evaluated by specialized psychologists, dietitians and therapists. Diabetes self-management education will be regularly exposed to patients
  Interventions: Other: type 1 diabetes structured education
- Conventional education group: Outpatients visit to endocrinologists when necessary in a conventional way.

INTERVENTIONS:
Other: type 1 diabetes structured education — The structured education is based on a regular outpatients visit.It is an education that integrated several diabetes related subjects,which mainly aimed at T1D self-management.
  Groups: Intensive structured education group

SUMMARY:
This study aims to clarify the underlying hereditary and autoimmune factors that contribute to clinical type 1 diabetes and gain a better understanding of the natural history of the disease.

ELIGIBILITY:
Inclusion Criteria:

1. diabetes diagnosed according to the report of WHO (World Health Organization) in 1999;
2. insulin dependence from disease onset,thus diagnosed with type 1 diabetes;
3. all patients gave informed consent to participate in the study and the protocol was approved by the Research Ethics Committee in second Xiangya hospital, Central South University.

Exclusion Criteria:

1. secondary diabetes mellitus;
2. pregnant women;
3. malignant disease.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: type 1 diabetes patients
Sampling Method: Probability Sample
Enrollment: 2110 (Actual)
Dates: Start 2016-10-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Effects of structured education on β-cell endocrine function progression of T1D patients. | Baseline and every three months afterwards.
  The natural progression of patients' β-cell endocrine functions was assessed by fasting C-peptide (FCP) and postprandial C-peptide (PCP) at each visit. FCP and PCP levels were measured at initial recruitment and every three months after that. The decay rate of β-cell endocrine function of patients in the two groups were compared.
  Serum C-peptide levels were measured by a chemiluminescence method using a commercial available kit (Adiva Centaur System, Siemens, Germany).

SECONDARY OUTCOMES:
Effects of structured education on blood sugar control. | Baseline and every three months afterwards.
  Patients' daily insulin dosage (U/Day) were collected at initial recruitment and each visit afterwards. And the above mentioned parameters in group 1(patients with structured education) and group2(patients without structured education) were compared.
Effects of structured education on blood sugar control. | Baseline and every three months afterwards.
  Patients' blood sugar levels were collected at initial recruitment and each visit afterwards. And the above mentioned parameters in group 1(patients with structured education) and group2(patients without structured education) were compared.
Effects of structured education on blood sugar control. | Baseline and every three months afterwards.
  Patients' HbA1c levels were collected at initial recruitment and each visit afterwards. And the above mentioned parameters in group 1(patients with structured education) and group2(patients without structured education) were compared.HbA1c concentration was tested by the Bio-Red Variant automatic measurement system.
Effects of structured education on metabolic control. | Baseline and every three months afterwards.
  Patients' body mass index (BMI) levels were collected at initial recruitment and each visit afterwards. And the above mentioned parameters in group 1(patients with structured education) and group2(patients without structured education) were compared.
Effects of structured education on metabolic control. | Baseline and every three months afterwards.
  Patients' systolic blood pressure (SBP) and diastolic blood pressure (DBP) levels were collected at initial recruitment and each visit afterwards. And the above mentioned parameters in group 1(patients with structured education) and group2(patients without structured education) were compared.
Effects of structured education on metabolic control. | Baseline and every three months afterwards.
  Patients' triglyceride (TG) and total cholesterol (TC) levels were collected at initial recruitment and each visit afterwards. And the above mentioned parameters in group 1(patients with structured education) and group2(patients without structured education) were compared.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Metabolism and Endocrinology, Second Xiangya Hospital, Central South University, Changsha, Hunan, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Deng C, Xie Y, Liu F, Tang X, Fan L, Yang X, Chen Y, Zhou Z, Li X. Simplified integration of optimal self-management behaviors is associated with improved HbA1c in patients with type 1 diabetes. J Endocrinol Invest. 2024 Nov;47(11):2691-2699. doi: 10.1007/s40618-024-02357-8. Epub 2024 Apr 11. PMID 38602658
- [Derived] Zhong T, Li X, Lei K, Tang R, Zhou Z, Zhao B, Li X. CXCL12-CXCR4 mediates CD57+ CD8+ T cell responses in the progression of type 1 diabetes. J Autoimmun. 2024 Feb;143:103171. doi: 10.1016/j.jaut.2024.103171. Epub 2024 Feb 1. PMID 38306953
- [Derived] Ji X, Zou W, Fan L, Zhou Z, Zhu X, Li X. Insulin resistance-related features are associated with cognitive decline: a cross-sectional study in adult patients with type 1 diabetes. Diabetol Metab Syndr. 2024 Jan 11;16(1):13. doi: 10.1186/s13098-023-01249-w. PMID 38212850
- [Derived] Huang F, Ji X, Xie Y, Li J, Li X, Zhou Z. Structured nutrition and advanced carbohydrate counting questionnaire for adult type 1 diabetes. Chin Med J (Engl). 2023 Jul 20;136(14):1753-1755. doi: 10.1097/CM9.0000000000002721. Epub 2023 Jun 1. No abstract available. PMID 37262038
- [Derived] Xie Y, Shi M, Ji X, Huang F, Fan L, Li X, Zhou Z. Insulin resistance is more frequent in type 1 diabetes patients with long disease duration. Diabetes Metab Res Rev. 2023 Sep;39(6):e3640. doi: 10.1002/dmrr.3640. Epub 2023 Apr 8. PMID 36964977
- [Derived] Chen Y, Xia Y, Xie Z, Zhong T, Tang R, Li X, Zhou Z. The Unfavorable Impact of DR9/DR9 Genotype on the Frequency and Quality of Partial Remission in Type 1 Diabetes. J Clin Endocrinol Metab. 2022 Jan 1;107(1):e293-e302. doi: 10.1210/clinem/dgab589. PMID 34390338
- [Derived] Zhu S, Liu F, Li J, Guan Y, Meng M, Li X, Zhou Z, Xu R, Li L. Development and validation of a self-management scale of type 1 diabetes for Chinese adults. J Int Med Res. 2020 Aug;48(8):300060520947588. doi: 10.1177/0300060520947588. PMID 32865059
- [Derived] Li X, Zhong T, Tang R, Wu C, Xie Y, Liu F, Zhou Z. PD-1 and PD-L1 Expression in Peripheral CD4/CD8+ T Cells Is Restored in the Partial Remission Phase in Type 1 Diabetes. J Clin Endocrinol Metab. 2020 Jun 1;105(6):dgaa130. doi: 10.1210/clinem/dgaa130. PMID 32236416
- [Derived] Xie Y, Liu F, Huang F, Lan C, Guo J, He J, Li L, Li X, Zhou Z. Establishment of a type 1 diabetes structured education programme suitable for Chinese patients: type 1 diabetes education in lifestyle and self adjustment (TELSA). BMC Endocr Disord. 2020 Mar 10;20(1):37. doi: 10.1186/s12902-020-0514-9. PMID 32151245